CLINICAL TRIAL: NCT07037836
Title: Inhaled Treprostinil (Tyvaso Nebulizer) For COPD Patients With Hypoxemia
Acronym: Tyvaso
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00118083
Record Dates: First submitted 2025-05-09; First posted 2025-06-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Hypoxemia
Keywords: Tyvaso; COPD; Hypoxemia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inhaled Treprostinil in COPD Patients With Hypoxemia and Preserved DLCO (Experimental)
  Interventions: Drug: Inhaled Treprostinil (Tyvaso Nebulizer)

INTERVENTIONS:
Drug: Inhaled Treprostinil (Tyvaso Nebulizer) — Participants will receive inhaled Treprostinil (Tyvaso nebulizer), 6 µg per breath, administered four times daily for 4 weeks. The starting dose will be 3 breaths per session. The dose will increase by 1 breath per session each week, as tolerated, to a target of 6 breaths per session by week 4. If adverse effects occur, participants will remain at the highest tolerated dose. The drug will be administered using the Tyvaso inhalation system provided by United Therapeutics. No changes to baseline COPD maintenance medications are allowed during the treatment period. Participants will be monitored for safety throughout the study.

SUMMARY:
The goal of this clinical trial is to evaluate whether inhaled Treprostinil (Tyvaso) can improve oxygen delivery and blood flow in the lungs in adults (age ≥40) with chronic obstructive pulmonary disease (COPD) and hypoxemia who have less severe reduction in lung blood volume (diffusing capacity of the lungs for carbon monoxide [DLCO] ≥45%).

The main questions it aims to answer are:

1. Does inhaled Treprostinil increase pulmonary capillary blood volume in ventilated lung regions, as measured by hyperpolarized xenon-129 magnetic resonance imaging (HP129Xe MRI)?
2. Does inhaled Treprostinil improve oxygen delivery (measured as red blood cell [RBC] chemical shift) and maintain or only slightly change pulmonary vascular resistance (measured by RBC oscillation amplitude)?
3. Can pre-treatment MRI parameters (RBC transfer and RBC oscillation amplitude) predict who will respond to inhaled Treprostinil?

Participants will:

* Use the Tyvaso nebulizer (inhaled Treprostinil) 4 times daily for 4 weeks, starting at 3 breaths per session and increasing to a maximum of 6 breaths per session as tolerated.
* Undergo HP129Xe MRI before and after treatment to assess regional lung function and oxygen exchange.
* Complete pulmonary function tests (PFTs), 6-minute walk tests (6MWT), and echocardiograms at the beginning and end of the study.
* Be monitored for adverse events, with a phone check-in midway through and after the treatment period.

DETAILED DESCRIPTION:
This is a single-arm, proof-of-concept study evaluating the effects of inhaled Treprostinil (Tyvaso nebulizer) on regional gas exchange and capillary blood oxygenation in patients with chronic obstructive pulmonary disease (COPD) and hypoxemia. The study will enroll 10 outpatient subjects aged ≥40 with a chronic bronchitis phenotype, confirmed COPD diagnosis, and a diffusing capacity of the lungs for carbon monoxide (DLCO) ≥45% predicted. All participants will receive inhaled Treprostinil via a 4-week dose titration protocol (starting at 3 breaths four times daily and increasing to 6 breaths as tolerated).

The primary objectives are to "determine the effects of inhaled Treprostinil on regional gas exchange and capillary blood oxygenation as measured by hyperpolarized xenon-129 magnetic resonance imaging (HP129Xe MRI), including ventilation defect percentage (VDP), membrane defect percentage, red blood cell (RBC) transfer defect percentage and normalized RBC oscillation amplitude and RBC frequency shift," and to "determine whether pre-treatment VDP, membrane defect percentage, RBC transfer defect percentage, RBC chemical shift and normalized RBC oscillation amplitude predict a positive response to inhaled Treprostinil."

Assessments will include HP129Xe MRI, spirometry with DLCO, 6-minute walk testing (6MWT), and echocardiography at baseline and after 4 weeks. Data will be analyzed for changes in regional lung function and oxygenation. Safety monitoring will focus on known adverse effects of inhaled Treprostinil including "cough, headache, hypotension, oropharyngeal pain, throat irritation and nausea," and will address more serious risks observed in the PERFECT trial (COPD exacerbation, respiratory failure, myocardial infarction, and death). By selecting subjects with DLCO ≥45% predicted and using a shorter 4-week treatment duration with titrated dosing, the study aims to mitigate these risks.

ELIGIBILITY:
Inclusion Criteria

* Outpatients of either gender, age ≥ 40.
* Clinical evidence of chronic bronchitis (a productive cough lasting more than 3 months within a 2-year period).
* Current or former cigarette smokers with a smoking history of 20 or more pack-years.
* Clinical diagnosis of chronic obstructive pulmonary disease (COPD) confirmed by spirometry demonstrating forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) ratio < 0.70, pre-bronchodilator FEV1 ≥ 30% predicted, and diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 45% predicted.
* On stable maintenance COPD medications including inhaled corticosteroids (ICS), long-acting beta agonists (LABA), long-acting muscarinic antagonists (LAMA), combination inhalers, azithromycin, or roflumilast (with no changes over the past 3 months).
* Patients with hypoxemia, evidenced by the use of supplemental oxygen at rest or during exercise (≤ 4 liters/minute).
* Willing and able to give informed consent and adhere to visit and protocol schedules (consent must be obtained prior to any study procedures).
* Women of childbearing potential must have a negative serum pregnancy test, confirmed prior to participation in this investigational protocol.

Exclusion Criteria

* Upper respiratory tract infection within 6 weeks (participants may be rescreened after this period).
* History of lung resection surgery or pleural decortication.
* Previous history of pneumothorax.
* Imaging evidence of interstitial lung disease, occupational lung disease, or chronic infectious lung disease.
* History of asthma.
* History of exposure to occupational or environmental hazards known to cause lung disease.
* Positive pregnancy test for women of childbearing potential.
* Major chronic illness that, in the judgment of the study physician, would interfere with participation in the study.

For Magnetic Resonance Imaging (MRI):

* Contraindications to MRI based on screening questionnaire responses.
* Participant is pregnant or lactating.
* Respiratory illness of bacterial or viral etiology within 6 weeks prior to MRI.
* Known cardiac arrhythmia.
* Participant does not fit into the hyperpolarized xenon-129 (^129Xe) vest coil used for MRI.
* Participant cannot hold their breath for 10 seconds.
* Participant is unlikely to comply with instructions during imaging.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percentage (VDP) on HP129XeMRI | Baseline and 4 weeks post-Tyvaso
  Defined as the region with ventilation signals < mean - 2SD, measured by HP129XeMRI and expressed as a percentage of total lung volume.
Membrane Defect Percentage on HP129XeMRI | Baseline and 4 weeks post-Tyvaso
  Defined as the region with membrane signals < mean - 2SD, measured by HP129XeMRI and expressed as a percentage of total lung volume.
Low Membrane Region Percentage on HP129XeMRI | Baseline and 4 weeks post-Tyvaso
  Defined as the region with membrane signals between 1SD and 2SD below the mean, measured by HP129XeMRI and expressed as a percentage of total lung volume.
RBC Transfer Defect Percentage on HP129XeMRI | Baseline and 4 weeks post-Tyvaso
  Defined as the region with RBC transfer signals < mean - 2SD, measured by HP129XeMRI and expressed as a percentage of total lung volume.
Low RBC Transfer Region Percentage on HP129XeMRI | Baseline and 4 weeks post-Tyvaso
  Defined as the region with RBC transfer signals between 1SD and 2SD below the mean, measured by HP129XeMRI and expressed as a percentage of total lung volume.
RBC Oscillation Amplitude Normalized for RBC Transfer Defect | Baseline and 4 weeks post-Tyvaso
  Measured using HP129XeMRI spectroscopy as a surrogate for pulmonary vascular resistance, normalized to RBC transfer signal intensity.
RBC Chemical Shift on HP129XeMRI Spectroscopy | Baseline and 4 weeks post-Tyvaso
  Frequency shift in RBC signal reflecting capillary blood oxygenation, measured using HP129XeMRI spectroscopy.

SECONDARY OUTCOMES:
Nadir SpO₂ During 6MWT | Baseline and 4 weeks post-Tyvaso treatment
  Lowest oxygen saturation (SpO₂) recorded during the 6-minute walk test, measured by pulse oximetry. The test is performed on room air unless SpO₂ drops below 89%, at which point supplemental oxygen is administered to maintain SpO₂ ≥89%.
Supplemental Oxygen Flow During 6MWT | Baseline and 4 weeks post-Tyvaso treatment
  Oxygen flow rate in liters per minute required to maintain SpO₂ ≥89% during the 6-minute walk test if room air is insufficient.
6-Minute Walk Distance (6MWD) | Baseline and 4 weeks post-Tyvaso treatment
  Total distance walked in meters during the 6-minute walk test, following ATS guidelines.
Dyspnea Score During 6MWT | Baseline and 4 weeks post-Tyvaso treatment
  Subjective rating of dyspnea severity on a 1-10 scale reported by participants at the end of the 6-minute walk test.
Peak Heart Rate (% Predicted) During 6MWT | Baseline and 4 weeks post-Tyvaso treatment
  Highest heart rate achieved during the 6-minute walk test, expressed as a percentage of predicted maximum heart rate.
Forced Expiratory Volume in 1 Second (FEV1) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  EV1 measured in liters and as a percentage of predicted value, assessed by spirometry.
Forced Vital Capacity (FVC) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  FVC measured in liters and as a percentage of predicted value, assessed by spirometry
Total Lung Capacity (TLC) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  TLC measured in liters and as a percentage of predicted value, assessed by lung volume testing.
Residual Volume (RV) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  RV measured in liters and as a percentage of predicted value, assessed by lung volume testing.
Diffusing Capacity for Carbon Monoxide (DLCO) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  DLCO measured in mL/min/mmHg and as a percentage of predicted value, assessed by single-breath method.
Carbon Monoxide Transfer Coefficient (KCO) - Absolute and % Predicted | Baseline and 4 weeks post-Tyvaso treatment
  KCO measured in mL CO/min/mmHg/L and as a percentage of predicted value, derived from DLCO and alveolar volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Asthma Allergy and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study. The consent form limits future data use to internal research on lung disease and COPD and does not authorize sharing of de-identified IPD with external investigators. Therefore, data cannot be made available to other researchers outside of the study team.